CLINICAL TRIAL: NCT07218276
Title: Passive Robots for Stroke Rehabilitation
Brief Title: Passive Robots for Stroke Rehabilitation: A Feasibility Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Chandramouli Krishnan, Principal Investigator, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: HUM00087962
Record Dates: First submitted 2025-10-15; First posted 2025-10-20 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Stroke
Keywords: synergy; upper extremity; stroke survivors; robot; hemiparesis; weakness
MeSH Terms: conditions — Stroke; Paresis; Asthenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Robotic Intervention (Experimental): Participants will receive upper extremity rehabilitation using SepaRRo and NeuRRoFES 2-5 times per week for 2-6 weeks
  Interventions: Device: Functional Training with SepaRRo and NeuRRoFES

INTERVENTIONS:
Device: Functional Training with SepaRRo and NeuRRoFES — Participants will perform functional movements (e.g., reach for targets) with their extremities. During movements, the devices will be used to assist or resist their motion. Participants may receive biofeedback of their movements to better engage them in training. Participants may receive assistance from the devices (including neuromuscular stimulation) and/or their less-impaired limb.

SUMMARY:
The purpose of this study is to examine the feasibility and effectiveness of a novel, multimodal approach that combines passive devices with noninvasive neuromuscular stimulation for upper extremity rehabilitation after stroke.

DETAILED DESCRIPTION:
About 800,000 individuals suffer from a stroke every year in the United States. The majority of stroke survivors often experience lingering deficits in upper extremity function. High-end robotic devices can improve outcomes and clinical productivity; however, these devices are expensive and bulky, making them not practical for many clinical or home environments. This study aims to evaluate the feasibility of low-cost non-motorized devices for stroke rehabilitation in a long-term intervention. The intervention will involve training with a table-top, semi-passive (i.e., no motors) exercise equipment called SepaRRo and commonly-used neuromuscular stimulation. The stimulation will be provided during functional activities using a custom controller (NeuRRoFES) to trigger stimulation. These instruments are designed to provide flexible, compliant assistance/resistance to improve upper extremity function and can be used in a home setting. The study will measure technical feasibility (e.g., qualitative survey, adherence, time on task, retention, ability to perform tasks) as well as clinical feasibility (i.e., changes in biomechanical, neurophysiological, and functional measures) of an intervention with these devices in stroke survivors. The findings aim to support the development of affordable, home-use rehabilitation systems for stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 75 years;
* Ischemic or hemorrhagic stroke confirmed by CT, MRI, or clinical criteria;
* No major deficits of sensation or proprioception;

Exclusion Criteria:

* Bilateral stroke
* Unable to think clearly and remember (Mini-Mental State Exam score < 22 and miniMOCA < 8);
* Uncontrolled Diabetes or Hypertension;
* Severe limitations of joint range of motion that will lead to inability of testing
* Severe spasticity and joint contractures that will lead to inability of testing
* Complete paresis with no possible movements
* Severe aphasia
* Any other medical condition that will significantly impact the study results
* Unable to obtain reliable motor evoked potentials
* Are pregnant or are actively trying to conceive
* Have a recent history of repeated fainting spells or syncope.
* Have a recent history of seizure (epilepsy) while on anti-seizure medication
* Have a recent history of skull fracture/head injury
* Have metal implants in the skull
* Have cardiac pacemakers

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2025-11-05 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Device Survey For Feasibility | Post-intervention (immediately following last session of intervention)
  Subjective feedback regarding feasibility of the device for training

OTHER OUTCOMES:
Retention | Post-intervention (immediately following last session of intervention)
  Measure of how many participants completed intervention
Adherence | Post-intervention (immediately following last session of intervention)
  Measure of percentage of sessions completed
Upper extremity Fugl-Meyer Score | Baseline and post-intervention measurements will be taken on separate days, within a week of the first and last sessions of the intervention, respectively.
  Changes in upper extremity Fugl-Meyer score from before the intervention (from baseline) to after its completion using publicly available scoring sheets. The Fugl-Meyer score is a measure of functional impairment and runs from 0 to 66 points, with higher numbers reflecting better outcome.
Reachable workspace | Baseline and post-intervention measurements will be taken on separate days, within a week of the first and last sessions of the intervention, respectively
  Changes in reachable workspace from before the intervention (from baseline) to after its completion). The reachable workspace area will be measured with SepaRRo obtained from optical encoders mounted in the device.
Voluntary hand opening | Baseline and post-intervention measurements will be taken on separate days, within a week of the first and last sessions of the intervention, respectively
  Changes in voluntary ability to open the hand from before the intervention (from baseline to after its completion). Voluntary hand opening will be measured with motion capture equipment.
Action Research Arm Test Score | Baseline and post-intervention measurements will be taken on separate days, within a week of the first and last sessions of the intervention, respectively
  Changes in the Action Research Arm Test Score from before the intervention (from baseline) to after its completion using publicly available scoring sheets. The Action Research Arm Test is a measure of arm functional ability and runs from 0 to 57 points, with higher numbers reflecting better outcome.
Box and Block (BBT) | Baseline and post-intervention measurements will be taken on separate days, within a week of the first and last sessions of the intervention, respectively
  Changes in functional measure of arm disability (BBT) from before the intervention (from baseline) to after its completion using publicly available scoring sheets.
Hand Strength | Baseline and post-intervention measurements will be taken on separate days, within a week of the first and last sessions of the intervention, respectively
  Changes in force produced by the hand from before the intervention (from baseline) to after its completion as measured by force production recorded with a dynamometer
Arm strength | Baseline and post-intervention measurements will be taken on separate days, within a week of the first and last sessions of the intervention, respectively
  Changes in force produced by the arm from before the intervention (from baseline) to after its completion as measured by force production recorded with a dynamometer
Muscle coordination | Baseline and post-intervention measurements will be taken on separate days, within a week of the first and last sessions of the intervention, respectively
  Changes in muscle coordination of the upper extremity muscles as measured using surface electromyography between before the intervention (from baseline) to after its completion.
Joint coordination | Baseline and post-intervention measurements will be taken on separate days, within a week of the first and last sessions of the intervention, respectively
  Changes in coordination of the upper extremity joints as measured motion capture between before the intervention (from baseline) to after its completion.
Corticospinal excitability | Baseline and post-intervention measurements will be taken on separate days, within a week of the first and last sessions of the intervention, respectively
  Changes in corticospinal excitability of the upper extremity muscles as measured using surface electromyography and transcranial magnetic stimulation between before the intervention (from baseline) to after its completion

CONTACTS AND LOCATIONS:
Overall Officials: Chandramouli Krishnan, PT, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan - NeuRRo Lab, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No